CLINICAL TRIAL: NCT02339259
Title: Rickettsial Disease in Febrile Hospitalised Patients in a Tertiary Referral Hospital in Bangladesh
Brief Title: Causes of Fever in Bangladeshi Patients
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Chittagong Medical College and Hospital (Other); University of Amsterdam (Other); Menzies School of Health Research (Other); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: BAKMAL1408
Record Dates: First submitted 2015-01-08; First posted 2015-01-15 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Rickettsial Disease
Keywords: Rickettsial disease; Febrile; Murine typhus; Scrub typhus; Diagnostic test; Clinical features
MeSH Terms: conditions — Rickettsia Infections; Fever; Typhus, Endemic Flea-Borne; Scrub Typhus | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, swab and crust specimen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Febrile patients: Febrile patients admitted to CMCH who have had malaria film and scrub typhus and murine typhus rapid test will be screened for enrolment.
  Interventions: Other: Observation
- Healthy: Healthy subjects with no recent history of fever will be recruited to provide control samples for the blood and plasma assays.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
Background:

The clinical features and prevalence of tropical rickettsial illnesses such as murine and scrub typhus in Bangladesh are unknown. Following testing for malaria, patients with undifferentiated fever are frequently treated empirically for typhoid or diagnosed clinically with a viral fever. Since murine and scrub typhus are common causes of fever in other countries in the region, it is likely they are prevalent in Bangladesh. Murine and scrub typhus may be treated cheaply and effectively with doxycycline.

Primary aim:

- Describe the clinical features of scrub and murine typhus in Bangladeshi patients

Secondary aims:

* Assess the proportion of patients screened for malaria having rickettsial illnesses
* Understand the pathophysiology of severe scrub typhus and murine typhus
* Prospective evaluation of rapid diagnostic tests for scrub and murine typhus

Methods:

Scrub typhus and murine typhus rapid tests will be introduced to CMCH in conjunction with existing malaria testing facilities. Consenting febrile adult patients who have had malaria and typhus rapid tests and meeting the entry criteria will be enrolled. Samples will be saved for serology and real time polymerase chain reaction (PCR) testing for O. tsutsugamushi and Rickettsia spp. A thorough history and examination will be undertaken. Hemodynamic status will be assessed by ultrasound upon enrolment. Patients will be followed up for outcome and a second sample will be taken for convalescent serological testing on day 14 where possible.

Analysis The proportion of patients screened for malaria with an acute febrile illness due to scrub typhus and murine typhus will be calculated. The clinical features of scrub and murine typhus, malaria and patients negative for these conditions will be compared. Healthy subject samples will be used to provide normal ranges. The sensitivity and specificity of the rapid tests will be assessed as compared to the gold standard of PCR and serology combined.

DETAILED DESCRIPTION:
Proposed activities:

The primary objective of this study are to assess the clinical features of patients with scrub or murine typhus infections presenting to CMCH. The proportion of cases screened for malaria and typhus who are diagnosed with scrub and murine typhus during the study period will be calculated, and the data made available for future empiric treatment guideline preparation.

Rapid antibody-based tests for scrub typhus and murine typhus will be made available for physicians to request alongside malaria testing in CMCH. Consenting febrile patients admitted to CMCH will be enrolled and history and clinical examination recorded. A sample will be taken for reference diagnostic testing at a later stage (including indirect fluorescent antibody (IFA) and real time PCR for scrub typhus and Rickettsia spp.)16. Samples will also be taken for testing of markers of pathophysiology (endothelial dysfunction neutrophil activation, cell death, cytokines). Where an eschar is found, the scab will be removed for real time-PCR. Where possible, patients will be invited back for a follow up 14 days after enrolment and a sample collected for paired serology assayed by IFA testing. Ultrasound based hemodynamic assessment will be performed to assess volume status and evidence of cardiac dysfunction.

The results of the ultrasound based hemodynamic assessment will be used to provide baseline information on patients with O. tsutsugamushi and Rickettsia spp. infection and other infections. This information may be used to plan further studies on the fluid management of these conditions.

Study design:

This is an observational study with no intervention. Febrile patients admitted to CMCH who have had malaria film and scrub typhus and murine typhus rapid test will be screened for enrolment. If patients meet the entry criteria, they will be enrolled after written informed consent has been given. Enrolled patients will then undergo study procedures (blood tests, physical examinations, follow-up).

Overall Description of study Participants:

The target population of this study is consenting adult patients who have had malaria and typhus rapid tests meeting the eligibility criteria admitted in CMCH. All study patients must meet the applicable inclusion and exclusion criteria.

During the study period, we aim to prospectively recruit consecutive patients until 300 patients are enrolled for whom there are paired admission and convalescent samples.

Data obtained from the malaria patients and patients without malaria or typhus will be used as comparator groups for the patients with typhus. The data from the 300 consecutive patients will be used to prospectively assess the sensitivity and specificity of the typhus diagnostic tests.

In addition, 30 healthy subjects with no recent history of fever will be recruited to provide control samples for the blood and plasma assays.

The total sample size is therefore estimated to be 330 (300 with paired serology and 30 healthy subjects).

ELIGIBILITY:
Patients

Inclusion Criteria:

1. Admitted to CMCH
2. Have had malaria and typhus rapid tests
3. Age≥12 years old
4. Febrile or history of fever for <3 weeks.
5. Written informed consent from patient or attending adult (for patient who lacks capacity) or parent (for those below 18)

Exclusion Criteria:

* Consent refused, or no adult (≥18 years) relative or guardian present to give consent in the case the patient lacks capacity to give consent.

Healthy subjects Inclusion

1. No known acute or chronic medical conditions
2. Asymptomatic
3. No febrile illness in the last 2 weeks
4. Age≥12 years old
5. Written informed consent from patient or parent (for those below 18)

Exclusion criteria:

1. Consent refused, or no adult (≥18 years) relative or guardian present to give consent in the case the patient is under 18 years.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is consenting adult patients who have had malaria and typhus rapid tests meeting the eligibility criteria admitted in CMCH. All study patients must meet the applicable inclusion and exclusion criteria.
  In addition, 30 healthy subjects with no recent history of fever will be recruited to provide control samples for the blood and plasma assays.
  The total sample size is therefore estimated to be 330 (300 patients with paired serology and 30 healthy subjects).
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The clinical features of severe and uncomplicated scrub typhus and murine typhus in Bangladeshi patients | 1 year

SECONDARY OUTCOMES:
Evaluation of markers of disease severity | 1 year
Hemodynamic status of patients with typhus | 1 year
Diagnostic accuracy of rapid diagnostic tests for scrub and murine typhus | 1 year
Proportion of acute rickettsial illnesses in patients screened for malaria | 1 year
Identification of vectors harbouring Rickettsia/Orientia spp. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hossain, Professor Md, Principal Investigator — Chittagong Medical College and Hospital
Locations (1):
- Chittagong Medical College Hosiptal, Chittagong, Bangladesh

REFERENCES:
- [Background] Suttinont C, Losuwanaluk K, Niwatayakul K, Hoontrakul S, Intaranongpai W, Silpasakorn S, Suwancharoen D, Panlar P, Saisongkorh W, Rolain JM, Raoult D, Suputtamongkol Y. Causes of acute, undifferentiated, febrile illness in rural Thailand: results of a prospective observational study. Ann Trop Med Parasitol. 2006 Jun;100(4):363-70. doi: 10.1179/136485906X112158. PMID 16762116
- [Background] Phongmany S, Rolain JM, Phetsouvanh R, Blacksell SD, Soukkhaseum V, Rasachack B, Phiasakha K, Soukkhaseum S, Frichithavong K, Chu V, Keolouangkhot V, Martinez-Aussel B, Chang K, Darasavath C, Rattanavong O, Sisouphone S, Mayxay M, Vidamaly S, Parola P, Thammavong C, Heuangvongsy M, Syhavong B, Raoult D, White NJ, Newton PN. Rickettsial infections and fever, Vientiane, Laos. Emerg Infect Dis. 2006 Feb;12(2):256-62. doi: 10.3201/eid1202.050900. PMID 16494751
- [Background] Miah MT, Rahman S, Sarker CN, Khan GK, Barman TK. Study on 40 cases of rickettsia. Mymensingh Med J. 2007 Jan;16(1):85-8. doi: 10.3329/mmj.v16i1.259. PMID 17344787
- [Background] Coleman RE, Monkanna T, Linthicum KJ, Strickman DA, Frances SP, Tanskul P, Kollars TM Jr, Inlao I, Watcharapichat P, Khlaimanee N, Phulsuksombati D, Sangjun N, Lerdthusnee K. Occurrence of Orientia tsutsugamushi in small mammals from Thailand. Am J Trop Med Hyg. 2003 Nov;69(5):519-24. PMID 14695089
- [Background] Tsay RW, Chang FY. Serious complications in scrub typhus. J Microbiol Immunol Infect. 1998 Dec;31(4):240-4. PMID 10496165
- [Background] Thap LC, Supanaranond W, Treeprasertsuk S, Kitvatanachai S, Chinprasatsak S, Phonrat B. Septic shock secondary to scrub typhus: characteristics and complications. Southeast Asian J Trop Med Public Health. 2002 Dec;33(4):780-6. PMID 12757226
- [Background] Sirisanthana V, Puthanakit T, Sirisanthana T. Epidemiologic, clinical and laboratory features of scrub typhus in thirty Thai children. Pediatr Infect Dis J. 2003 Apr;22(4):341-5. doi: 10.1097/01.inf.0000059400.23448.57. PMID 12690274
- [Background] Kim DM, Chung JH, Yun NR, Kim SW, Lee JY, Han MA, Lee YB. Scrub typhus meningitis or meningoencephalitis. Am J Trop Med Hyg. 2013 Dec;89(6):1206-11. doi: 10.4269/ajtmh.13-0224. Epub 2013 Oct 28. PMID 24166036
- [Background] Kim DM, Kim SW, Choi SH, Yun NR. Clinical and laboratory findings associated with severe scrub typhus. BMC Infect Dis. 2010 Apr 30;10:108. doi: 10.1186/1471-2334-10-108. PMID 20433689
- [Background] LEVINE HD. Pathologic study of thirty-one cases of scrub typhus fever with especial reference to the cardiovascular system. Am Heart J. 1946 Mar;31:314-28. doi: 10.1016/0002-8703(46)90313-4. No abstract available. PMID 21018737
- [Background] Paris DH, Phetsouvanh R, Tanganuchitcharnchai A, Jones M, Jenjaroen K, Vongsouvath M, Ferguson DP, Blacksell SD, Newton PN, Day NP, Turner GD.
- [Background] Paris DH, Phetsouvanh R, Tanganuchitcharnchai A, Jones M, Jenjaroen K, Vongsouvath M, Ferguson DP, Blacksell SD, Newton PN, Day NP, Turner GD. Orientia tsutsugamushi in human scrub typhus eschars shows tropism for dendritic cells and monocytes rather than endothelium. PLoS Negl Trop Dis. 2012 Jan;6(1):e1466. doi: 10.1371/journal.pntd.0001466. Epub 2012 Jan 10. PMID 22253938
- [Background] Moron CG, Popov VL, Feng HM, Wear D, Walker DH. Identification of the target cells of Orientia tsutsugamushi in human cases of scrub typhus. Mod Pathol. 2001 Aug;14(8):752-9. doi: 10.1038/modpathol.3880385. PMID 11504834
- [Background] Gillespie JJ, Ammerman NC, Beier-Sexton M, Sobral BS, Azad AF. Louse- and flea-borne rickettsioses: biological and genomic analyses. Vet Res. 2009 Mar-Apr;40(2):12. doi: 10.1051/vetres:2008050. Epub 2008 Nov 28. PMID 19036234
- [Background] Civen R, Ngo V. Murine typhus: an unrecognized suburban vectorborne disease. Clin Infect Dis. 2008 Mar 15;46(6):913-8. doi: 10.1086/527443. PMID 18260783
- [Background] Rovery C, Brouqui P, Raoult D. Questions on Mediterranean spotted fever a century after its discovery. Emerg Infect Dis. 2008 Sep;14(9):1360-7. doi: 10.3201/eid1409.071133. PMID 18760001
- [Background] Watthanaworawit W, Turner P, Turner C, Tanganuchitcharnchai A, Richards AL, Bourzac KM, Blacksell SD, Nosten F. A prospective evaluation of real-time PCR assays for the detection of Orientia tsutsugamushi and Rickettsia spp. for early diagnosis of rickettsial infections during the acute phase of undifferentiated febrile illness. Am J Trop Med Hyg. 2013 Aug;89(2):308-310. doi: 10.4269/ajtmh.12-0600. Epub 2013 Jun 3. PMID 23732256
- [Background] Blacksell SD, Bryant NJ, Paris DH, Doust JA, Sakoda Y, Day NP. Scrub typhus serologic testing with the indirect immunofluorescence method as a diagnostic gold standard: a lack of consensus leads to a lot of confusion. Clin Infect Dis. 2007 Feb 1;44(3):391-401. doi: 10.1086/510585. Epub 2007 Jan 3. PMID 17205447
- [Background] Jiang J, Chan TC, Temenak JJ, Dasch GA, Ching WM, Richards AL. Development of a quantitative real-time polymerase chain reaction assay specific for Orientia tsutsugamushi. Am J Trop Med Hyg. 2004 Apr;70(4):351-6. PMID 15100446
- [Background] Henry KM, Jiang J, Rozmajzl PJ, Azad AF, Macaluso KR, Richards AL. Development of quantitative real-time PCR assays to detect Rickettsia typhi and Rickettsia felis, the causative agents of murine typhus and flea-borne spotted fever. Mol Cell Probes. 2007 Feb;21(1):17-23. doi: 10.1016/j.mcp.2006.06.002. Epub 2006 Jul 1. PMID 16893625